CLINICAL TRIAL: NCT03579251
Title: An Intervention to Increase Retention in Care Among HIV-Positive Black Men
Brief Title: Black Men's Care, and Intervention to Re-Engage HIV+ Black Men in Care
Acronym: BMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1K23MH111402-01A1 (NIH); 1K23MH111402-01A1 (NIH)
Record Dates: First submitted 2018-05-03; First posted 2018-07-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: 1) Semi-structured, qualitative interviews; 2) protocol development; 3) single-arm pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilot test (Other): 12 weeks of behavioral intervention (Black Men's Care), including an in-person session and two-way SMS, with a three-month follow-up period post-intervention.
  Interventions: Behavioral: Black Men's Care

INTERVENTIONS:
Behavioral: Black Men's Care — 12 weeks of behavioral intervention, including an in-person session and two-way SMS, to re-engage in HIV care HIV-positive Black men who have fallen out of care

SUMMARY:
The proposed study aims to develop an intervention that is strategic in that it will 1) be a focused on an approach that combines an in-person session with post-session, two-way text messaging to continue the intervention and reinforce the gains from the in-person session and 2) ultimately find HIV+ Black men who have sex with men who have left HIV care where they are likely to present (e.g., city and county health clinics, community-based organizations, emergency rooms).

DETAILED DESCRIPTION:
The overarching goal of this application is to develop and conduct a preliminary test of a "portable" intervention, "Black Men's Care" (BMC), to re-engage in HIV care HIV+ Black men who have sex with men who have left HIV care (+BMSM-LC) that is flexible with respect to where it can be conducted. The aims of the study are: Aim 1-to conduct formative research to develop BMC content and optimize its delivery; Aim 2-to develop BMC, a theory-based, combination in-person and text messaging (mHealth) intervention for +BMSM-LC; and Aim 3-to evaluate the acceptability, feasibility, and preliminary outcomes of BMC in preparation for submitting an R01 proposal to finalize and conduct an efficacy trial of BMC. Aims 1 and 2 will comprise the formative phase of the proposed study. Aim 1 will consist of semi-structured interviews with 2 staff members at each of 3 city and county health clinics, 3 community-based organizations, and 3 emergency rooms to identify effective settings for intervention. Aim 2 will consist of semi-structured interviews with 10 +BMSM-LC and 10 HIV+ Black men who have sex with men who remain in care to develop intervention content. Findings from these semi-structured interviews and Aim 1 will be used to develop a preliminary intervention protocol that will be refined across 2 sets of 3 sequential, single-subject iterations of the intervention sampled by age (n=3 for ages 18 to 29 years, n =3 for ages 30 and up). For Aim 3, a pilot study of 18 +BMSM-LC purposively sampled by age will assess acceptability, feasibility, and preliminary outcomes of BMC for re-engaging +BMSM-LC in care. The research and career development activities of this K23 proposal will allow the PI to achieve the goal of becoming an independent, R01-funded investigator. The PI will gain a broad range of critical skills (e.g., intervention development; qualitative research methods; trial design, safety monitoring, and process and outcome evaluation) and experiences to address the health needs of vulnerable populations at greatest risk of morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Staff (interviews): administrators and frontline workers who have worked in their respective positions for at least 6 months and have a caseload that includes +BMSM or a position at an organization that serves +BMSM. These staff members will be recruited from the San Francisco Bay Area.
* HIV-positive Black male patients (interviews): 1) HIV+, 2) self-identified as men who have sex with men, 3) 18 years or older, 4) have left HIV care, as indicated by less than 2 appointment in the past year and no scheduled appointments in the next 6 months or are engaged in care, as indicated by at least 2 appointment at least 90 days apart in the last year, and 5) live in or near the San Francisco Bay Area
* HIV-positive Black male patients (pilot study): 1) HIV+, 2) self-identified as men who have sex with men, 3) 18 years or older, 4) have left HIV care, as indicated by less than 2 appointment in the past year and no scheduled appointments in the next 6 months, 5) live in or near the San Francisco Bay Area, and 6) must also be available for the Pre-Intervention Survey; the BMC in-person session, 12 weeks of SMS, and Post-Intervention Survey upon completion of the intervention; and 3-Month Follow-Up after the intervention

Exclusion Criteria:

* Non-native English speaker

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A man living with HIV from a population that is disparately affect by HIV, particularly men who have sex with men.
Enrollment: 28 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Level of Engagement in Care--Appointments in the Past Six Months | At baseline, at the end of the intervention (at three months), and three months after the intervention (at six months)
  This is a simple, explicit behavioral outcome measure. The measures is to ask participants whether they have attended HIV care appointment in the past 6 months (response options: yes or no)
Change from Baseline Level of Engagement in Care--Future Appointments | At baseline, at the end of the intervention (at three months), and three months after the intervention (at six months)
  This is a simple, explicit behavioral outcome measure. The measures is to ask participants whether they have a future HIV care appointment schedule (response options: yes or no)

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire--8-item version | At 12 weeks (at three months)
  The measure assesses participants' satisfaction with the intervention. Response options range from 1 (a lower degree of satisfaction) to 4 (a higher degree of satisfaction), and the mean of the eight items will be calculated to yield an overall score. Higher values indicated greater satisfaction.
Number of Missed Appointments | At six months (i.e., at three-month follow-up after the three-month intervention)
  This measure is contingent upon whether patient and provider consent to give access to the medical record. This is a measure of the number of schedule appointments missed during a six-month period.
CD4 Count | At six months (i.e., at three-month follow-up after the three-month intervention)
  This measure is contingent upon whether patient and provider consent to give access to the medical record. This is the last measure of the patient's CD4 count.
Viral Load | At six months (i.e., at three-month follow-up after the three-month intervention)
  This measure is contingent upon whether patient and provider consent to give access to the medical record. This is the viral load number or, if applicable, if the viral load is "undetectable."
Percent of Appointments Missed | At six months (i.e., at three-month follow-up after the three-month intervention)
  This measure is contingent upon whether patient and provider consent to give access to the medical record. This is the ratio of the number of schedule appointments missed to the number of scheduled appointments during a six-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Vincent, Ph.D., MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States